CLINICAL TRIAL: NCT06356948
Title: The Effect of Tranexamic Acid Rate of Administration on Blood Pressure in Healthy Pregnant Women Scheduled for Elective Cesarean Delivery Under Spinal Anesthesia - A Prospective, Randomized, Double-blind, Non-inferiority Trial.
Brief Title: Rate of Tranexamic Acid Administration on Blood Pressure (RateTXA) Study.
Acronym: RateTXA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H23-02918
Record Dates: First submitted 2024-03-18; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Healthy Participants
Keywords: tranexamic acid; infusion rate; post-partum hemorrhage; hypotension; cesarean delivery
MeSH Terms: conditions — Postpartum Hemorrhage; Hypotension | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double-blind, non-inferiority trial.
  Arm 1: Intravenous infusion of TXA 1g (10 mL) administered over 1 minute. Arm 2: Intravenous infusion of TXA 1g (10 mL) administered over 10 minutes
Who Masked: Participant, Care Provider, Investigator
Masking Description: An anesthesiologist or anesthesia assistant not involved in the study will draw up TXA and labelling them based on the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rapid-rate administration of TXA (Active Comparator): This group will be administered tranexamic acid over 1 minute
  Interventions: Drug: Tranexamic Acid (TXA)
- Slow-rate administration of TXA (Active Comparator): This group will be administered tranexamic acid over 10 minutes
  Interventions: Drug: Tranexamic Acid (TXA)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — Study drug administration
  Other Names: Tranexamic Acid

SUMMARY:
Tranexamic acid is a well-established treatment for post-partum hemorrhage. This study aims to examine the effect of tranexamic acid administration rates on blood pressure changes over 1 minute compared to 10 minutes in healthy pregnant patients scheduled for cesarean delivery.

DETAILED DESCRIPTION:
Women who are clinically diagnosed with post-partum hemorrhage during a vaginal or cesarean delivery should be immediately administered tranexamic acid according to the World Health Organization's recommendation. Tranexamic acid is a drug that inhibits the breakdown of fibrin clots which reduces blood loss. However, due to the risk of hypotension, the product monograph for TXA advises against rapid intravenous (IV) administration. Other clinical studies have also reported an increased incidence of nausea, vomiting, and visual disturbances; nonetheless, the results of these trials suggest that these side effects may be related to properties of TXA rather than the rate of administration. Therefore, the investigators of this study aim to determine if the rate of tranexamic acid administration has an effect on blood pressure in healthy pregnant patients who are scheduled for cesarean delivery under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients ≥34 weeks gestational age, for elective cesarean delivery under single-shot spinal anesthesia.
* American Society of Anesthesiologists (ASA) Physical Status Class 2.
* Patients ≥19 years of age.

Exclusion Criteria:

* Known history of pre-existing hypertension or hypertension disorders of pregnancy.
* Having recently taken a medication to treat high blood pressure (e.g. labetolol, hydralazine, nifedipine)
* Having recently taken a medication that could alter blood pressure, which could include beta those prescribed for anxiety (e.g. propranolol) or sedative pre-medication (e.g. midazolam, lorazepam).
* Known allergic reaction or hypersensitivity to TXA or any other TXA homologue.
* Elective cesarean delivery requiring general anesthesia or a neuraxial technique other than a single-shot spinal (e.g. Epidural or Combined Spinal Epidural).
* Patients who are unable to give informed consent due to a language barrier as the study team only speaks English and will be unable to complete consent process and study procedure appropriately.
* Patients arriving late to the surgical day care with <90 min prior to scheduled cesarean delivery time resulting in potential delay for the operating room or inadequate time for consent and full execution of the protocol.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure from baseline over 15 minutes post-TXA administration between groups. | 15 minutes starting from the time of completed TXA administration.
  Change in systolic blood pressure from baseline over 15 minutes post-TXA administration between study and control groups

SECONDARY OUTCOMES:
Incidence of nausea | Up to 4 hours from time of TXA administration until time of discharge from the recovery room
  sensation of self-reported nausea documented every 5 minutes.
Incidence of vomiting | Up to 4 hours from time of TXA administration until time of discharge from the recovery room
  vomiting documented every 5 minutes.
Incidence of hypotension | Up to 4 hours from time of TXA administration until time of discharge from the recovery room
  Incidence of systolic blood pressure reduction greater than or equal to 20% of baseline
Incidence of hypertension | Up to 4 hours from time of TXA administration until time of discharge from the recovery room
  Incidence of systolic blood pressure elevation greater than or equal to 20% of baseline
Incidence of central nervous system side effects | Up to 4 hours from time of TXA administration until time of discharge from the recovery room
  composite outcome of neurologic side effects including dizziness, headache, visual disturbances (photopsia) or facial flushing. These measures will be self-reported and documented every 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — Department of Anesthesia BC Women's Hospital
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sentilhes L, Winer N, Azria E, Senat MV, Le Ray C, Vardon D, Perrotin F, Desbriere R, Fuchs F, Kayem G, Ducarme G, Doret-Dion M, Huissoud C, Bohec C, Deruelle P, Darsonval A, Chretien JM, Seco A, Daniel V, Deneux-Tharaux C; Groupe de Recherche en Obstetrique et Gynecologie. Tranexamic Acid for the Prevention of Blood Loss after Vaginal Delivery. N Engl J Med. 2018 Aug 23;379(8):731-742. doi: 10.1056/NEJMoa1800942. PMID 30134136
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Boisselle ME, Zaphiratos VV, Fortier A, Richebe P, Loubert C. Comparison of carbetocin as a bolus or an infusion with prophylactic phenylephrine on maternal heart rate during Cesarean delivery under spinal anesthesia: a double-blinded randomized controlled trial. Can J Anaesth. 2022 Jun;69(6):715-725. doi: 10.1007/s12630-022-02227-y. Epub 2022 Mar 30. PMID 35352277
- [Background] Cheema HA, Ahmad AB, Ehsan M, Shahid A, Ayyan M, Azeem S, Hussain A, Shahid A, Nashwan AJ, Mikus M, Lagana AS. Tranexamic acid for the prevention of blood loss after cesarean section: an updated systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol MFM. 2023 Aug;5(8):101049. doi: 10.1016/j.ajogmf.2023.101049. Epub 2023 Jun 11. PMID 37311484
- [Background] Abdel-Aleem H, Alhusaini TK, Abdel-Aleem MA, Menoufy M, Gulmezoglu AM. Effectiveness of tranexamic acid on blood loss in patients undergoing elective cesarean section: randomized clinical trial. J Matern Fetal Neonatal Med. 2013 Nov;26(17):1705-9. doi: 10.3109/14767058.2013.794210. Epub 2013 May 10. PMID 23574458
- [Background] Novikova N, Hofmeyr GJ, Cluver C. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2015 Jun 16;2015(6):CD007872. doi: 10.1002/14651858.CD007872.pub3. PMID 26079202
- [Background] Pacheco LD, Clifton RG, Saade GR, Weiner SJ, Parry S, Thorp JM Jr, Longo M, Salazar A, Dalton W, Tita ATN, Gyamfi-Bannerman C, Chauhan SP, Metz TD, Rood K, Rouse DJ, Bailit JL, Grobman WA, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Tranexamic Acid to Prevent Obstetrical Hemorrhage after Cesarean Delivery. N Engl J Med. 2023 Apr 13;388(15):1365-1375. doi: 10.1056/NEJMoa2207419. PMID 37043652
- [Background] Sentilhes L, Senat MV, Le Lous M, Winer N, Rozenberg P, Kayem G, Verspyck E, Fuchs F, Azria E, Gallot D, Korb D, Desbriere R, Le Ray C, Chauleur C, de Marcillac F, Perrotin F, Parant O, Salomon LJ, Gauchotte E, Bretelle F, Sananes N, Bohec C, Mottet N, Legendre G, Letouzey V, Haddad B, Vardon D, Madar H, Mattuizzi A, Daniel V, Regueme S, Roussillon C, Benard A, Georget A, Darsonval A, Deneux-Tharaux C; Groupe de Recherche en Obstetrique et Gynecologie. Tranexamic Acid for the Prevention of Blood Loss after Cesarean Delivery. N Engl J Med. 2021 Apr 29;384(17):1623-1634. doi: 10.1056/NEJMoa2028788. PMID 33913639
- [Background] Vogel JP, Oladapo OT, Dowswell T, Gulmezoglu AM. Updated WHO recommendation on intravenous tranexamic acid for the treatment of post-partum haemorrhage. Lancet Glob Health. 2018 Jan;6(1):e18-e19. doi: 10.1016/S2214-109X(17)30428-X. Epub 2017 Oct 31. No abstract available. PMID 29100880
- [Background] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Ng W, Jerath A, Wasowicz M. Tranexamic acid: a clinical review. Anaesthesiol Intensive Ther. 2015;47(4):339-50. doi: 10.5603/AIT.a2015.0011. Epub 2015 Mar 23. PMID 25797505
- [Background] McCormack PL. Tranexamic acid: a review of its use in the treatment of hyperfibrinolysis. Drugs. 2012 Mar 26;72(5):585-617. doi: 10.2165/11209070-000000000-00000. PMID 22397329